CLINICAL TRIAL: NCT04391361
Title: The Safety and Effectiveness of Cholinergic Receptor Block Therapy in the Treatment of Amyotrophic Lateral Sclerosis
Brief Title: The Safety and Effectiveness of Cholinergic Receptor Block Therapy in the Treatment of ALS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: lj11128
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Amyotrophic Lateral Sclerosis; Respiratory Function; Scopolamine
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Respiratory Aspiration | interventions — Scopolamine; Atropine; Edaravone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial group (Experimental)
  Interventions: Drug: Scopolamine, atropine, edaravone and dexmedetomidine
- control group (Placebo Comparator)
  Interventions: Drug: Edaravone

INTERVENTIONS:
Drug: Scopolamine, atropine, edaravone and dexmedetomidine — The patients were treated with scopolamine, atropine, edaravone and dexmedetomidine dissolved in saline.
  Arms: trial group
Drug: Edaravone — The patients was treated with edaravone dissolved in the same volume of saline as the intervention applied in the experimental group.
  Arms: control group

SUMMARY:
Thirty cases of amyotrophic lateral sclerosis patients were recruited from the neurology department of Ruijin Hospital, the pain department and the encephalopathy center of Luwan Branch of Ruijin Hospital. After the informed consent was signed, they were divided into a trial group and a control group. Each group contains 15 cases. The patients in the control group was treated with edaravone dissolved in saline during hospitalization, while the patients in the trial group was treated with edaravone, scopolamine, atropine and dexmedetomidine. Both groups of subjects were treated for 7 days within 3 weeks, followed by a buffer period of 3 weeks for observation, which was one treatment course. The total treatment protocol contains 3 treatment courses (or 18 weeks). Patients with amyotrophic lateral sclerosis were evaluated before treatment and 6, 12, 18, 24, 36, 48 weeks after treatment. The observations include whether the functional scores of patients with amyotrophic lateral sclerosis, Norris amyotrophic lateral sclerosis score, amyotrophic lateral sclerosis self-score, forced expiratory volume in one second, partial pressure of oxygen and maximum displacement of the hyoid were superior to those before treatment, and whether the partial pressure of carbon dioxide was inferior to those before treatment. Study hypothesis: Cholinergic receptor blocking therapy for amyotrophic lateral sclerosis is safe and effective in improving motor function and delaying disease progression in patients with amyotrophic lateral sclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should voluntarily participate in the experiment by signing an informed consent form.
2. Patients should comply with the research process and cooperate with the interventions applied throughout the experiment.
3. Patients should be between 30 and 65 years of age, and both sexes are acceptable.
4. Patients should comply with the diagnostic criteria and exclusion criteria for amyotrophic lateral sclerosis in the Chinese Guidelines for the Diagnosis and Treatment of Amyotrophic Lateral Sclerosis developed by the Chinese Society of Neurology of the Chinese Medical Association in 2012.
5. Patient's amyotrophic lateral sclerosis history must not exceed 5 years.
6. ALS functional scale score (ALSFRS-R) should be ≥ 2 points for each patients.

Exclusion Criteria:

1. Patients with cardiac conduction block, severe ventricular insufficiency, severe hepatorenal insufficiency and severe, progressive or uncontrolled major organ and systemic disease.
2. High or low blood pressure: systolic blood pressure >150 or <110 mmHg; bradycardia (<60 beats per minute).
3. Patients with ventilator-assisted ventilation.
4. Patients who are allergic to research intervention drugs.
5. Patients with obvious signs of dementia.
6. Female patients who are pregnant or breastfeeding or who have a plan to become pregnant in the near future.
7. Persons with other psychiatric disorders that may affect the assessment of their condition.
8. Severely obese patients (BMI >35kg/m2).

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Effective | 48 weeks
  Forced expiratory volume in one second (FVC%) or ALS functional rating scale score (ALSFR, minimum score: 0, maximum score: 48, higher score is related to a better outcome) was elevated.
Ineffective | 48 weeks
  Forced expiratory volume in one second (FVC%) or ALS functional rating scale score (ALSFR, minimum score: 0, maximum score: 48, higher score is related to a better outcome) was decreased or remained unchanged.

SECONDARY OUTCOMES:
Effective | 48 weeks
  Partial pressure of oxygen (PO2), maximum displacement of the hyoid or the modified Norris scale score (minimum score: 0, maximum score: 100, higher score is related to a better outcome) was elevated or partial pressure of carbon dioxide (PCO2) was decreased or remained unchanged.
Ineffective | 48 weeks
  Partial pressure of carbon dioxide (PCO2) was elevated, or partial pressure of oxygen (PO2), maximum displacement of the hyoid or the modified Norris scale score (minimum score: 0, maximum score: 100, higher score is related to a better outcome) was decreased or remained unchanged.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Liu, Professor, Study Chair — Department of Neurology, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Department of neurology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) was available to other researchers.